CLINICAL TRIAL: NCT02099357
Title: Creatine or Vitamin D Supplementation in Persons With Spinal Cord Injury Undergoing Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Samuel Amorim, Bsc, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FADEUPAFA20132015
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Creatine; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Daily supplementation with 3g of dextrose during eight weeks and placebo ampoules each two weeks.
  Interventions: Dietary Supplement: Placebo
- Creatine (Experimental): Daily supplementation with 3g of monohydrate creatine during eight weeks. Placebo ampoules each two weeks.
  Interventions: Dietary Supplement: Creatine
- Vitamin D (Active Comparator): Daily supplementation with 3g of dextrose during eight weeks. Vitamin D supplementation, 25000 IU each two weeks.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Creatine — Daily supplementation with 3g of monohydrate creatine during 8 weeks
  Arms: Creatine
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Vitamin D — Vitamin D supplementation with 25000 IU each two weeks during eight weeks
  Arms: Vitamin D

SUMMARY:
The purpose of this study is to determine the effects of creatine monohydrate or vitamin D supplementation on strength gains following a traditional resistance training program for adults with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury
* Minimum time since injury: 3 months

Exclusion Criteria:

* Participation in resistance training programmes in the previous 6 months
* Creatine or vitamin D supplementation in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 8 weeks
Sum of 4 skinfold | 8 weeks
  Triceps, Biceps, Subscapular and Iliac crest
Corrected Arm Muscle Area | 8 weeks
Seated Medicinal Ball Throw | 8 weeks
Handgrip Strength with Hand Dynamometer | 8 weeks
Manual Wheelchair Slalom Test | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vitor H Teixeira, PhD, Study Director — Faculdade de Ciências da Nutrição e Alimentação, Universidade do Porto; Rui Corredeira, PhD, Study Chair — Faculdade de Desporto, Universidade do Porto; Samuel Amorim, Bsc, Principal Investigator — Faculdade de Desporto, Universidade do Porto
Locations (2):
- Portugal (2):
  - Centro de Medicina de Reabilitação da Região Centro - Rovisco Pais, Cantanhede, Coimbra District
  - Centro de Reabilitação do Norte, Vila Nova de Gaia, Porto District